CLINICAL TRIAL: NCT06292819
Title: Effects of Photobiomodulation on Insomnia in the Elderly: Clinical Trials of Phototherapy Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wan-Ju Cheng, Doctor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC2-214
Record Dates: First submitted 2024-02-17; First posted 2024-03-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Photobiomodulation
Keywords: rhythm; light therapy; insomnia; sleep; older
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright light (Active Comparator)
  Interventions: Device: Bright light
- Near-infrared light (Active Comparator)
  Interventions: Device: Near-infrared light
- Bright light+ near-infrared light (Active Comparator)
  Interventions: Device: Bright light+ near-infrared light

INTERVENTIONS:
Device: Bright light — Bright light will use a 5000-10,000 Lux LED light source. Exposure is for 60 minutes daily, between 7pm and 9pm.
  Arms: Bright light
Device: Near-infrared light — Near-infrared light will use a wavelength of 850nm and a dose range of 1 - 6.5 joules/cm2. It is fixed on the neck with a band, the light source contacts the back of the neck, and is used for 60 minutes before going to bed.
  Arms: Near-infrared light
Device: Bright light+ near-infrared light — After using the bright light device, then use the near-infrared light device on the back of the neck before going to bed.
  Arms: Bright light+ near-infrared light

SUMMARY:
The study will recruit 60 participants aged 60 and above, who suffered from insomnia for at least 3 months. Sleep parameters and chronotypes assessed with questionnaires and actigraphy, daytime sleepiness, and biological rhythm (dim light melatonin onset) will be measured. The intervention involves light exposure using a prototype device developed by GCSOL Tech Co., Ltd., a company with expertise in light therapy research and development. Three conditions will be tested (1) bright light; (2) near-infrared light; (3) bright light+ near-infrared light. Data analysis will employ paired t-tests to compare sleep parameters and dim light melatonin onset before and after treatment. Kruskal-Wallis tests and multivariate linear regression will be used to examine differences between intervention groups, controlling for gender and age. Safety analysis will include monitoring adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pittsburgh Sleep Quality Index score is 8 or above.
* Early wakening ( 30 minutes before expected), or interruptted sleep for more than 30 minutes, lasting for more than 3 months.

Exclusion Criteria:

* Movement disorder, inability to move independently.
* Skin diseases, skin cancer, photosensitive skin diseases, or taking drugs that may cause photosensitivity (lithium salts, melatonin, antibiotics, A acid).
* Eye diseases such as glaucoma, diabetic retinopathy, and cataracts.
* Bipolar disorder.
* Light-induced epilepsy.
* Sleep disorders such as sleep apnea and involuntary leg twitching.
* Currently taking sedative-hypnotic drugs or receiving other non-drug treatments.
* Beck depression inventory-II score is greater than 13 points.
* Those who use cardiac rhythm regulators or artificial cardiopulmonary pacemakers.
* Acute illness.
* Abnormal blood pressure or fever.
* Pregnancy and pregnant women.
* Special physical abnormalities and sensory nerve abnormalities.
* Infectious diseases.
* Coagulation disorder.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Actigraphy-derived sleep indicators | Baseline and the third week.
  Participants will continue to wear activity recording watches during the three weeks of the study. We will capture weekly average sleep duration, sleep onset latency, wake time after falling asleep, and sleep efficiency.
Dim-light melatonin onset | Baseline and the third week.
  Participants will be required to provide saliva samples for melatonin analysis within their home environment. These samples will be collected at 30-minute intervals starting from 18:00 and continuing until 1 hour after their habitual sleep time on both the initial and final study dates. The concentration of salivary melatonin will be assessed utilizing a direct melatonin enzyme-linked immunosorbent assay (ELISA) kit. The Dim Light Melatonin Onset (DLMO) will be determined using the two standard deviation threshold method, which involves calculating the average of the first three melatonin data points and then adding two standard deviations to this average.
Sleep quality | Baseline and the third week.
  Pittsburgh Sleep Quality Index (PSQI) ranges from 0 (better) to 21 (worse).
Emotional state | Baseline and the third week.
  Beck Depression Inventory-II ranges from 0 (better) to 63 (worse).

SECONDARY OUTCOMES:
Daytime sleepiness | Baseline and the third week.
  Epworth Sleepiness Scale ranges from 0 (better) to 24 (worse).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No